CLINICAL TRIAL: NCT05287191
Title: MAGNesium and Digoxin Versus AMiodarone for Fast Atrial Fibrillation in the ICU (MAGNAM Trial)
Brief Title: MAGNAM Trial, Magnesium Versus Amiodarone in Atrial Fibrillation in Critical Care
Acronym: MAGNAM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3664
Record Dates: First submitted 2022-01-06; First posted 2022-03-18 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation New Onset
Keywords: Atrial fibrillation; critical illness
MeSH Terms: conditions — Atrial Fibrillation; Critical Illness | interventions — Magnesium Sulfate; Amiodarone

STUDY DESIGN:
Intervention Model Description: Individual patient, pragmatic, comparative effectiveness, randomised, controlled trial
Who Masked: Outcomes Assessor
Masking Description: Blinded follow up for key outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Intravenous magnesium sulphate as first line followed by digoxin IV loading as second line and then amiodarone IV as third line treatments for fast Atrial Fibrillation
  Interventions: Drug: Magnesium sulfate and then Digoxin
- Standard of care arm (Active Comparator): Intravenous amiodarone as compactor group intervention
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Magnesium sulfate and then Digoxin — We will test MgSO4 and then digoxin IV (in 3 divided dose) as second line therapy with amiodarone IV as third line. Digoxin will be protocolised to commence between 30 minutes and 12 hours after MgSO4 if fast Atrial Fibrillation persists as initially designated (dose 1). Undiluted IV digoxin (12 mcg/kg) will be administered in 3 divided doses (6, 3 and 3 mcg/kg) separated by approximately 6 hrs (i.e. dose 1 at 30 mins - 12 hours after MgSO4, followed by dose 2 at -6 hrs and dose 3 at the approximately 12 hrs). Patients with renal dysfunction (creatinine clearance <60 ml/min measured by the Modification of diet in renal disease formula) will receive a reduced dose of 8 mcg/kg in 3 divided doses (4, 2, and 2 mcg/kg) separated by the same time intervals. In the trial intervention group, amiodarone will be given approximately 120 mins after digoxin if necessary whilst completing the digoxin dose. Amiodarone as a 150 mg infusion over 10 minutes followed by 900 mg over 24 hours.
  Arms: Experimental arm
Drug: Amiodarone — We will test Amiodarone (150mg IV then 900mg IV over the next 24 hours ) as first line treatment in the standard of care group. No more than 2g MgSO4 be delivered over 2 hours maximum for this group in the first 24 hours after randomisation unless clinically indicated for measured hypomagnesaemia (a value below the index hospital laboratories lower limit of normal).
  Arms: Standard of care arm

SUMMARY:
A multi-centre, non-blinded, comparative effectiveness, randomised controlled trial. Patients will be prospectively enrolled from Critical Care Units and will be assessed for study enrollment based on inclusion/exclusion criteria at the time of the onset of fast atrial fibrillation (AF)(irregular and often rapid heart rate). The authors hypothesize that high dose Magnesium Sulphate with the addition of Digoxin as a second line treatment will improve the success rate in returning the heart to normal rhythm as well as speed of resolution of critical illness in new onset rapid atrial fibrillation in the critically ill cared for in general ICUs.

DETAILED DESCRIPTION:
This is a Multi-centre, randomised controlled, clinical trial that is comparing a Stepwise Strategy of Magnesium Followed by Digoxin, With an Amiodarone Backup vs a Strategy of First-line Amiodarone to See Which is More Effective in Returning the Heart to Normal Rhythm After Experiencing Rapid Atrial Fibrillation in General ICUs. It will take place in Critical Care Units in Toronto Health Sciences Centres over a course of 2 years. The sample size is 200 patients.

Investigational Product and Planned Use Magnesium sulphate

The trial intervention will be Magnesium sulphate followed by digoxin as second line therapy with Amiodarone as third line. The Standard of care intervention will be Amiodarone as first line treatment in the and then no more than 2g MgSO4 be delivered.

Data will be collected retrospectively at the outcome timepoints.

Statistical Analysis:

This analysis will be conducted using the intention to treat principle, therefore all randomised patients will be included in the main analysis. Crossovers and protocol violations will remain in their original study group.

Baseline data will be summarized per group for continuous variables using means and standard deviations or medians and interquartile ranges as indicated the distribution and for discrete variables using frequencies and percentages. For the rate / rhythm co-primary outcome the authors will use a sentinel time point analysis at the 6 and 24 hour time points assuming there no / very low competing risk for death using a multivariate regression model to test for differences between groups and adjusting for baseline variables such as age, hospital site, shock status (requirement for inotropes Y/N), mechanical ventilation (Y/N) and known chronic atrial fibrillation. For the ICU length of stay co-primary outcome the authors recognise the competing risk of death and for this outcome and the authors propose to use Fine and Gray models adjusting for the stratification variables (as above). Estimates will be presented as sub-distribution hazards and 95% confidence intervals. The authors will test for interaction between sub-group and treatment and present the estimates per sub-group.

All secondary outcomes are binary and differences between groups will be tested using Chi square test or Fisher exact test as appropriate. Missing data will be uncommon for our key outcome data considering the nature of this data. The authors do not propose to use imputation for missing data in these primary or secondary analyses.

ELIGIBILITY:
Inclusion Criteria: Each participant must meet all of the following inclusion criteria to participate in this study:

1. Admitted to a participating hospital ICU
2. A newly documented episode of fast Atrial Fibrillation with heart rate >120/min confirmed by a 12-lead ECG assessment regardless of baseline rhythm (note- The AF can be acute or chronic diagnosis)
3. Undergoing, or able to commence continuous electrocardiographic monitoring ("telemetry") as part of their routine clinical care
4. Treating physician determines the patient has clinically significant AF that requires medical treatment

Exclusion Criteria:

1. Age <18 years
2. Palliative goals of care or expected to die in the next 12 hours
3. Fast Atrial Fibrillation (>120/min) present for > 48 hours
4. Treatment with digoxin or a class I or III anti-arrhythmic medication within the preceding 24 hours
5. MgSO4 dose of > 3g IV in the last 2 hours.
6. History of high grade Atrio-Ventricular conduction block or bradyarrhythmia without pacemaker
7. Non-cardiac indication or contraindication to one of the study treatments (hypertensive disorders of pregnancy, pre-term labour, neuromuscular junction disorders i.e. known Myasthenia gravis; documented prior history of amiodarone toxicity or relative contraindication such as thyroid disease, cirrhosis, pulmonary fibrosis, etc.)
8. Recent cardiac surgery during index hospital admission
9. Known pregnancy
10. Sustained (more than 10 continuous seconds documented on a rhythm strip) ventricular arrhythmia within the past 24 hours
11. Known or suspected pre-excitation syndrome
12. Persistent hyperkalemia > 6mmol/l despite treatment
13. Previously enrolled in the MAGNAM trial
14. Recent lung transplantation (during this admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate control (<110 beats per minute) and/or restoration of normal sinus | 6 hours
  heart rate control
ICU free days | 90 days
  ICU free days

SECONDARY OUTCOMES:
Hospital mortality | Up to 90 days
  Hospital mortality
Heart rate | 24 hours
  Maintenance rate control
Continuation of trial intervention | Up to 90 days
  Continuation of any of the drugs in the intervention (magnesium, digoxin or amiodarone) at the time of discharge from ICU
Presence of new rate and / or rhythm control medications at the time of first ICU discharge | Up to 90 days
  Presence of new rate and / or rhythm control medications
Serious adverse events | Up to 90 days
  Serious adverse events
Avoidance of amiodarone | Up to 90 days
  Avoidance of amiodarone during the ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Brian H Cuthbertson, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (5):
- Canada (5):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Blinded data will be shared with other researchers after verification of their study plan and discussion about recognitions
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after publication
Access Criteria: Contact PI